CLINICAL TRIAL: NCT04722978
Title: Standard Chemotherapy Plus Moxifloxacin as First-line Treatment for Metastatic Triple-negative Breast Cancer : a Multicenter, Double-blind, Placebo-controlled, Phase 3 Trial
Brief Title: Standard Chemotherapy Plus Moxifloxacin as First-line Treatment for Metastatic Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSUCC-003
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Gemcitabine; Carboplatin; Anti-Bacterial Agents; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Gemcitabine combined with carboplatin plus moxifloxacin or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Gemcitabine combined with carboplatin plus moxifloxacin
  Interventions: Drug: Gemcitabine and carboplatin plus antibiotic (moxifloxacin)
- Control group (Placebo Comparator): Gemcitabine combined with carboplatin plus placebo
  Interventions: Drug: Gemcitabine combined with carboplatin plus placebo

INTERVENTIONS:
Drug: Gemcitabine and carboplatin plus antibiotic (moxifloxacin) — Standard chemotherapy (gemcitabine and carboplatin) plus antibiotic (moxifloxacin)
  Other Names: Gemcitabine 1000mg/m^2 IV on days 1 and 8; cycled every 21 days Carboplatin AUC 2 IV on days 1 and 8; cycled every 21 days Moxifloxacin 0.4 PO once daily days 1-5; cycled every 21 days
  Arms: Experimental group
Drug: Gemcitabine combined with carboplatin plus placebo — Standard chemotherapy (gemcitabine and carboplatin) plus placebo
  Other Names: Gemcitabine 1000mg/m^2 IV on days 1 and 8; cycled every 21 days Carboplatin AUC 2 IV on days 1 and 8; cycled every 21 days Placebo 0.4 PO once daily days 1-5; cycled every 21 days
  Arms: Control group

SUMMARY:
The primary objective of this study is to compare progression-free survival (PFS) of patients with metastatic triple-negative breast cancer randomised to treatment with standard chemotherapy plus moxifloxacin or placebo.

DETAILED DESCRIPTION:
This is a multicenter, randomised, double-blind, placebo-controlled, phase 3 trial. The main purposes of this study are to examine the efficacy and safety of standard chemotherapy plus moxifloxacin or placebo as first-line treatment in patients with metastatic triple-negative breast cancer. This study is designed to recruit up to 228 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) score of 0 to 1.
* Histologically confirmed invasive ductal carcinoma, no specific type (NOS)
* ER negative and progesterone receptor (PR) negative (defined as < 1% positive cells by IHC), human epidermal growth factor receptor 2 (HER2) negative (defined as IHC 0-1 staining or fluorescent in situ hybridization (FISH) negative).
* No prior therapy after first recurrence or diagnosis of metastatic disease.
* At least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Neutrophil-to-lymphocyte ratios (NLR) in peripheral blood ≥ 2.
* Adequate organ function including bone marrow, renal function, hepatic function, and cardiac reserve (Left ventricular ejection fraction (LVEF) by echocardiogram ≥45%).
* Compliance with the study protocol.
* Have provided written and signed informed consent.

Exclusion Criteria:

* Pregnant or breast feeding.
* Definitive breast cancer susceptibility gene (BRCA) mutation, Programmed Cell Death-Ligand 1 (PD-L1) positive, microsatellite instability-high (MSI-H), and mismatch repair deficient (dMMR).
* Patients who are receiving or will receive other biological agents or immunotherapy.
* Uncontrolled medical problems.
* Evidence of active acute or chronic infection.
* Hepatic, renal, cardiac, or bone marrow dysfunction as detailed above.
* Concurrent malignancy or history of other malignancy within the last five years.
* Known severe hypersensitivity to moxifloxacin
* Patients were unable or unwilling to comply with program requirements.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 36 months
  The interval from the date of randomization until the first date on which progression, or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-yu Yuan, M.D., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China